CLINICAL TRIAL: NCT00467649
Title: A Phase 4, Randomized, Open Label, Parallel Group, Multicenter Study to Characterize Regimens of Basal Insulin Intensified With Either Symlin® or Rapid Acting Insulin in Patients With Type 2 Diabetes
Brief Title: A Study to Characterize Regimens of Basal Insulin Intensified With Either Symlin® or Rapid Acting Insulin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACA401
Record Dates: First submitted 2007-04-27; First posted 2007-05-01 (Estimated); Results first posted 2009-06-04 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Symlin; Amylin; insulin; Humalog; Novolog; Apidra
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — pramlintide; Insulin, Short-Acting; Insulin Lispro; Insulin Aspart; insulin glulisine; Insulin Glargine; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: pramlintide acetate (Symlin); Drug: basal insulin (Lantus® [insulin glargine], or Levemir® [insulin detemir])
- Group B (Active Comparator)
  Interventions: Drug: rapid acting insulin (Humalog® [insulin lispro], Novolog® [insulin aspart], or Apidra® [insulin glulisine]); Drug: basal insulin (Lantus® [insulin glargine], or Levemir® [insulin detemir])

INTERVENTIONS:
Drug: pramlintide acetate (Symlin) — subcutaneous injection (60 mcg or 120 mcg), immediately prior to major meals
  Other Names: Symlin
  Arms: Group A
Drug: rapid acting insulin (Humalog® [insulin lispro], Novolog® [insulin aspart], or Apidra® [insulin glulisine]) — subcutaneous injection, dosing based on titration guidelines
  Arms: Group B
Drug: basal insulin (Lantus® [insulin glargine], or Levemir® [insulin detemir]) — subcutaneous injection, dosing based on titration guidelines

SUMMARY:
This will be a randomized, open label, parallel group, multicenter study. There will be two phases in the study. Phase 1 (Baseline to Week 24) will compare the efficacy and safety of regimens of basal insulin intensified with either Symlin or rapid acting insulin in patients with type 2 diabetes who have either been on a prior regimen of insulin for less than 6 months and were taking less than 50 U total of insulin per day OR are candidates for the initiation of insulin therapy. The purpose of Phase 2 (Week 24 to Week 36) is to explore further intensification of diabetes regimens in patients failing to achieve HbA1c <=6.5% at Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Has a clinical diagnosis of type 2 diabetes mellitus
* Has an HbA1c >7.0% and ≤10.0%
* Has a BMI of ≥25 kg/m^2 and ≤50 kg/m^2
* Has been on a regimen of insulin for less than 6 months and is taking less than 50 U total of insulin per day, OR has not been on a pre existing insulin regimen and is a candidate for the initiation of basal insulin therapy

Exclusion Criteria:

* Has experienced recurrent severe hypoglycemia requiring assistance during the past 6 months
* Requires the use of drugs that stimulate gastrointestinal motility
* Has been previously treated with Symlin (or has participated in a Symlin clinical study)
* Is currently being treated with any of the following medications: *Over-the-counter antiobesity agents (including, but not limited to, herbal supplements) or prescription antiobesity agents (including orlistat [Xenical®] and sibutramine [Meridia®]); *Oral, intravenous, or intramuscular systemic steroids by oral or potent inhaled or intrapulmonary steroids that are known to have a high rate of systemic absorption; *Drugs that directly affect gastrointestinal motility, including but not limited to: dopamine antagonists (e.g., metoclopramide [Reglan®]), opiates or anticholinergics; and chronic (more than 10 days within a 6-month period) macrolide antibiotics such as erythromycin and newer derivatives; *Investigational medications
* Has a history or presence of any of the following: *Eating disorders (including anorexia and/or bulimia); *Bariatric surgery (gastric bypass, gastric banding, or gastroplasty)
* Is currently enrolled in a weight-loss program or plans to enroll in a weight-loss program before termination of the study
* Has donated blood within 30 days of study start or plans to donate blood during the duration of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2007-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (37):
- United States (37):
  - Research Site, Northport, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Loma Linda, California
  - Research Site, Aurora, Colorado
  - Research Site, Hollywood, Florida
  - Research Site, Maitland, Florida
  - Research Site, Miami, Florida
  - Research Site, North Miami Beach, Florida
  - Research Site, Plantation, Florida
  - Research Site, Roswell, Georgia
  - Research Site, Peoria, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Jackson, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Butte, Montana
  - Research Site, Las Vegas, Nevada
  - Research Site, Hamilton, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Albany, New York
  - Research Site, Staten Island, New York
  - Research Site, Mentor, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Bridgeville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Aiken, South Carolina
  - Research Site, Bartlett, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Olympia, Washington
  - Research Site, Spokane, Washington

REFERENCES:
- [Derived] Peyrot M, Rubin RR, Polonsky WH, Best JH. Patient reported outcomes in adults with type 2 diabetes on basal insulin randomized to addition of mealtime pramlintide or rapid-acting insulin analogs. Curr Med Res Opin. 2010 May;26(5):1047-54. doi: 10.1185/03007991003634759. PMID 20199136

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A (Phase 1 SYMLIN): SYMLIN treatment (120 mcg prior to major meals) was initiated on Day 1. Basal insulin was titrated throughout the study
- Group B (Phase 1 RA Insulin): Rapid acting insulin (RA Insulin: variable dosing, titrated to optimize postprandial glucose control) was initiated at Week 4. Basal insulin was titrated throughout the study
- Group C (Phase 2 SYMLIN): Patients from Group A, who achieved HbA1c goal at Week 24, continued Phase 1 treatment during Phase 2
- Group D (Phase 2 SYMLIN+RA): Patients from Group A, who did not achieve HbA1c goal at Week 24, continued Phase 1 treatment and initiated RA insulin during Phase 2
- Group E (Phase 2 RA Insulin): Patients from Group B, who achieved HbA1c goal at Week 24, continued Phase 1 treatment during Phase 2
- Group F (Phase 2 RA Insulin + SYMLIN): Patients from Group B, who did not achieve HbA1c goal at Week 24, continued Phase 1 treatment and initiated SYMLIN during Phase 2
Period: Phase 1 (Randomized Population)
Arm/Group | Group A (Phase 1 SYMLIN) | Group B (Phase 1 RA Insulin) | Group C (Phase 2 SYMLIN) | Group D (Phase 2 SYMLIN+RA) | Group E (Phase 2 RA Insulin) | Group F (Phase 2 RA Insulin + SYMLIN)
Started | 57 (One patient randomized to the SYMLIN group withdrew consent prior to receiving the first dose) | 56 | 0 | 0 | 0 | 0
Intent to Treat | 56 | 56 | 0 | 0 | 0 | 0
Completed | 48 | 50 | 0 | 0 | 0 | 0
Not Completed | 9 | 6 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator Decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 4 | 0 | 0 | 0 | 0
Not completed — Withdrawal of Consent | 4 | 2 | 0 | 0 | 0 | 0
Period: Phase 2 (Intent-to-Treat Population)
Arm/Group | Group A (Phase 1 SYMLIN) | Group B (Phase 1 RA Insulin) | Group C (Phase 2 SYMLIN) | Group D (Phase 2 SYMLIN+RA) | Group E (Phase 2 RA Insulin) | Group F (Phase 2 RA Insulin + SYMLIN)
Started | 0 | 0 | 17 | 31 | 14 | 36
Completed | 0 | 0 | 17 | 29 | 14 | 35
Not Completed | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal of Consent | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Phase 1 SYMLIN) | Group B (Phase 1 RA Insulin) | Total
Number analyzed (Participants) | 56 | 56 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 49 | 95
  >=65 years | 10 | 7 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (11.35) | 53.6 (9.70) | 54.3 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 34 | 37 | 71
Region of Enrollment [Number; unit: participants]
  United States | 56 | 56 | 112
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 155.1 (39.60) | 164.3 (49.61) | 159.7 (44.92)
Fasting Serum Lipids [Mean (Standard Deviation); unit: mg/dL]
  Total Cholesterol | 167.53 (47.054) | 169.86 (49.121) | 168.70 (47.903)
  HDL | 44.71 (11.893) | 41.77 (9.468) | 43.23 (10.790)
  LDL | 89.15 (38.386) | 90.41 (34.114) | 89.78 (36.133)
  Triglycerides | 174.13 (108.257) | 193.59 (159.508) | 183.95 (136.273)
HbA1c [Mean (Standard Deviation); unit: Percent] | 8.19 (0.840) | 8.25 (0.816) | 8.22 (0.825)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 116.31 (15.427) | 117.15 (13.198) | 116.73 (14.297)
Weight [Mean (Standard Deviation); unit: kg] | 107.87 (21.893) | 103.46 (17.908) | 105.67 (20.032)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients Achieving HbA1c <=7% at Week 24 With no Gain in Body Weight From Baseline and no Incidence of Severe Hypoglycemia
Description: A severe hypoglycemia is defined as an event during which the patient required the assistance of another individual (including aid in ingestion of oral carbohydrate); and/or required the administration of glucagon injection, intravenous glucose, or other medical intervention.
Time Frame: 24 Weeks
Population: Phase 1 Intent-to-Treat LOCF. LOCF: If a treated patient has missing result value at week 24, then last observed value before week 24 and after baseline is carried forward to impute the week 24 value.
Measure: Number; unit: Percent
Arm/Group | Group A (Phase 1 SYMLIN) | Group B (Phase 1 RA Insulin)
Number analyzed (Participants) | 56 | 56
Percent | 30.4 | 10.7
Statistical Analysis 1: Comparison: Group A (Phase 1 SYMLIN) vs Group B (Phase 1 RA Insulin); Test type: Superiority or Other; p = 0.0180, Fisher Exact

2. Secondary Outcome: Percentage of Patients Achieving HbA1c <=7% at Week 24
Description: This is a component of the primary endpoint
Time Frame: 24 Weeks
Population: Phase 1 Intent-to-Treat
Measure: Number; unit: Percent
Arm/Group | Group A (Phase 1 SYMLIN) | Group B (Phase 1 RA Insulin)
Number analyzed (Participants) | 56 | 56
Percent | 44.6 | 55.4

3. Secondary Outcome: Percentage of Patients With no Weight Gain at Week 24
Description: This is a component of the primary endpoint
Time Frame: 24 Weeks
Population: Phase 1 Intent-to-Treat
Measure: Number; unit: Percent
Arm/Group | Group A (Phase 1 SYMLIN) | Group B (Phase 1 RA Insulin)
Number analyzed (Participants) | 56 | 56
Percent | 46.4 | 14.3

4. Secondary Outcome: Percentage of Patients With a Severe Hypoglycemia Adverse Event
Description: This is a component of the primary endpoint.
Time Frame: 24 Weeks
Population: Phase 1 Intent-to-Treat
Measure: Number; unit: Percent
Arm/Group | Group A (Phase 1 SYMLIN) | Group B (Phase 1 RA Insulin)
Number analyzed (Participants) | 56 | 56
Percent | 0.0 | 0.0

5. Secondary Outcome: Change in HbA1c From Baseline at Week 24
Description: Baseline values are presented in the Baseline Characteristics section
Time Frame: From Baseline to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Group A (Phase 1 SYMLIN) | Group B (Phase 1 RA Insulin)
Number analyzed (Participants) | 56 | 56
Percent | -1.11 (0.17) | -1.27 (0.17)

6. Secondary Outcome: Change in Body Weight From Baseline at Week 24
Description: Baseline values are presented in the Baseline Characteristics section
Time Frame: From Baseline to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Group A (Phase 1 SYMLIN) | Group B (Phase 1 RA Insulin)
Number analyzed (Participants) | 56 | 56
kg | 0.02 (0.68) | 4.65 (0.68)

7. Secondary Outcome: Change in Waist Circumference From Baseline at Week 24
Description: Baseline values are presented in the Baseline Characteristics section
Time Frame: From Baseline to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Group A (Phase 1 SYMLIN) | Group B (Phase 1 RA Insulin)
Number analyzed (Participants) | 53 | 56
cm | -0.63 (0.87) | 2.17 (0.86)

8. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline at Week 24
Description: Baseline values are presented in the Baseline Characteristics section
Time Frame: From Baseline to Week 24
Population: Phase 1 Intent-to-Treat
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Group A (Phase 1 SYMLIN) | Group B (Phase 1 RA Insulin)
Number analyzed (Participants) | 45 | 50
mg/dL | -29.0 (7.32) | -37.8 (7.69)

9. Secondary Outcome: Fasting Serum Lipids Change From Baseline to Week 24
Time Frame: Baseline, week 24
Population: Phase 1 Intent-to-Treat
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Group A (Phase 1 SYMLIN) | Group B (Phase 1 RA Insulin)
Number analyzed (Participants) | 47 | 49
mg/dL
  Total Cholesterol | -1.81 (5.826) | 5.27 (4.649)
  HDL | 1.11 (1.190) | 1.65 (1.075)
  LDL | 2.36 (4.456) | 9.12 (3.865)
  Triglycerides | -28.96 (12.442) | -31.98 (13.883)

10. Secondary Outcome: Phase 2: Change in HbA1c at Week 36
Description: Two changes are calculated, the first by subtracting Week 36 value from the Phase 1 Baseline value (total change over 36 weeks), the second by subtracting the Week 36 value from the Phase 2 Baseline value (change from week 24 to week 36 only).
Time Frame: Phase 1 Baseline, Phase 2 Baseline at Week 24, Week 36
Population: Phase 2 Intent-to-Treat
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Group C (Phase 2 SYMLIN) | Group D (Phase 2 SYMLIN+RA) | Group E (Phase 2 RA Insulin) | Group F (Phase 2 RA Insulin + SYMLIN)
Number analyzed (Participants) | 17 | 30 | 14 | 36
Percent
  Phase 1 Baseline | 8.35 (0.214) | 8.03 (0.140) | 7.85 (0.183) | 8.38 (0.145)
  Change From Phase 1 Baseline to Week 36 | -1.96 (0.238) | -0.68 (0.174) | -1.49 (0.189) | -0.99 (0.157)
  Phase 2 Baseline at Week 24 | 6.26 (0.121) | 7.57 (0.171) | 6.14 (0.107) | 7.32 (0.170)
  Change From Phase 2 Baseline to Week 36 | 0.14 (0.062) | -0.23 (0.123) | 0.22 (0.097) | 0.07 (0.113)

11. Secondary Outcome: Phase 2: Change in Body Weight at Week 36
Description: as for outcome 10
Time Frame: Phase 1 Baseline, Phase 2 Baseline at Week 24, Week 36
Population: Phase 2 Intent-to-Treat
Measure: Mean (Standard Error); unit: kg
Arm/Group | Group C (Phase 2 SYMLIN) | Group D (Phase 2 SYMLIN+RA) | Group E (Phase 2 RA Insulin) | Group F (Phase 2 RA Insulin + SYMLIN)
Number analyzed (Participants) | 17 | 30 | 14 | 36
kg
  Phase 1 Baseline | 109.98 (4.916) | 104.83 (3.959) | 104.42 (7.341) | 105.30 (2.210)
  Change From Phase 1 Baseline to Week 36 | -0.80 (2.096) | 1.34 (0.933) | 3.90 (1.488) | 4.51 (0.761)
  Phase 2 Baseline at Week 24 | 108.50 (5.656) | 105.67 (4.045) | 107.87 (7.801) | 110.68 (2.507)
  Change From Phase 2 Baseline to Week 36 | 0.69 (0.654) | 0.50 (0.303) | 0.44 (0.518) | -0.86 (0.353)

12. Other Pre Specified Outcome: Hypoglycemia Adverse Events
Description: MILD: patient reported symptoms consistent with hypoglycemia that may or may not have been documented by glucose monitoring at the time of symptoms. Symptoms did not greatly interrupt or interfere with the patients daily activities. Symptoms dissipated spontaneously or upon eating.
  MODERATE: Patient reported symptoms consistent with hypoglycemia that may or may not have been documented by glucose monitoring at the time of symptoms. Symptoms interrupted or interfered with the patients daily activities and required immediate self treatment (e.g. carbohydrate ingestion).
  SEVERE: Patient required the assistance of another individual (including aid in ingestion of oral carbohydrate): and/or required the administration of glucagon injection, intravenous glucose, or other medical intervention.
Time Frame: 36 weeks
Measure: Number; unit: participants
Arm/Group | Group A (Phase 1 SYMLIN) | Group B (Phase 1 RA Insulin) | Group C (Phase 2 SYMLIN) | Group D (Phase 2 SYMLIN+RA) | Group E (Phase 2 RA Insulin) | Group F (Phase 2 RA Insulin + SYMLIN)
Number analyzed (Participants) | 56 | 56 | 17 | 31 | 14 | 36
participants
  Mild | 31 | 46 | 7 | 18 | 9 | 19
  Moderate | 12 | 13 | 0 | 1 | 2 | 3
  Severe | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Group A (Phase 1 SYMLIN) | Group B (Phase 1 RA Insulin) | Group C (Phase 2 SYMLIN) | Group D (Phase 2 SYMLIN+RA) | Group E (Phase 2 RA Insulin) | Group F (Phase 2 RA Insulin + SYMLIN)
Serious Adverse Events (participants affected / at risk) | 1/56 | 5/56 | 0/17 | 0/31 | 0/14 | 0/36
Other Adverse Events (participants affected / at risk) | 29/56 | 28/56 | 9/17 | 11/31 | 4/14 | 11/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Phase 1 SYMLIN) (N=56) | Group B (Phase 1 RA Insulin) (N=56) | Group C (Phase 2 SYMLIN) (N=17) | Group D (Phase 2 SYMLIN+RA) (N=31) | Group E (Phase 2 RA Insulin) (N=14) | Group F (Phase 2 RA Insulin + SYMLIN) (N=36)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Phase 1 SYMLIN) (N=56) | Group B (Phase 1 RA Insulin) (N=56) | Group C (Phase 2 SYMLIN) (N=17) | Group D (Phase 2 SYMLIN+RA) (N=31) | Group E (Phase 2 RA Insulin) (N=14) | Group F (Phase 2 RA Insulin + SYMLIN) (N=36)
Nausea (Gastrointestinal disorders) | 12 (16) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 5 (5) | 1 (1) | 2 (2) | 1 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (11) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 5 (5) | 0 (0) | 2 (3) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less